CLINICAL TRIAL: NCT04019301
Title: Caring for Caregivers With Mind-body Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Houston (Other)
Collaborators: Brigham and Women's Hospital (Other); Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34AT010081 (NIH)
Record Dates: First submitted 2019-06-21; First posted 2019-07-15 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Caregiver Distress; Physical Function; Quality of Life
Keywords: Cancer Caregiver; Qigong; Feasibility; Caregiver distress

STUDY DESIGN:
Intervention Model Description: Cancer caregivers will be randomized to one of three conditions: (1) a community-based qigong program; (2) an internet-based qigong program; or (3) a self-care control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Community-based Qigong Group (Experimental): Participants randomized into this group follow one, 75 minutes class per week supplemented by home practice for 20 minutes on 3 additional days.
  Interventions: Other: Baduanjin Qigong, Community-based
- Internet-based Qigong Group (Experimental): Participants randomized into this group follow two online sessions for 40 minutes each, also supplemented by home practice for 20 minutes on 3 additional days.
  Interventions: Other: Baduanjin Qigong, Internet-based
- Self-Care Control Group (No Intervention): The Self-care control group, will be requested not to practice any Qigong during the study. Participants will be provided with an educational book on caregiving that includes self-guided activities related to caregiving and caregiver health (The Caregiver Helpbook: Powerful Tools for Caregiving). The book's evidence-based program is designed to provide caregivers the tools to increase their self-care and their confidence to handle difficult situations, emotions, and decisions. In addition, study staff will call participants in the self-care control group once a month.

INTERVENTIONS:
Other: Baduanjin Qigong, Community-based — The Community-based Qigong group, will attend one 75 minute long Qigong class per week for 12 weeks. Additionally, participants practice Qigong at home for 20 minutes a day, 3 days a week. Printed materials will be provided to guide home practice.
  Other Names: Eight Brocades Regimen
  Arms: Community-based Qigong Group
Other: Baduanjin Qigong, Internet-based — The Internet-guided Qigong group will be given a computer tablet to access online Qigong classes. All participants assigned to this group will be provided with a tutorial to use the Qigong program by the research coordinator. Participants will be asked to follow a 40 minute long Qigong class twice a week for 12 weeks, and to practice an additional 20 minutes a day, 3 days a week. All sessions will be completed at home.
  Other Names: Eight Brocades Regimen
  Arms: Internet-based Qigong Group

SUMMARY:
This pilot study will lay the foundation for the first large-scale trial evaluating the psychosocial and physical health benefits of a widely available and promising Qigong intervention (Eight Brocades) for distressed cancer caregivers (CCGs). CCGs represent a well-defined, large and growing subset of a larger population of CGs that overlap greatly in the constellations of morbidities that lead to high levels of distress. The multi-modal nature of the Eight Brocades Qigong regimen explicitly targets both psychosocial and physical functional symptoms, thus expanding the scope of mind-body studies for CGs to date, which have largely focused on stress management and psychological well-being. This pilot study, and the eventual large-scale comparative effectiveness trial, explores the effectiveness of Qigong training delivered in both community-based group classes and through self-guided internet-based modules supplemented with one-on-one virtual learning support. This trial will be the first to explore the delivery of Qigong to caregivers using an internet-based program, potentially leading to wider accessibility to mind-body therapies, and providing an alternative to community-based group-class learning.

DETAILED DESCRIPTION:
Caregivers (CGs) often experience significant psychological and physical distress leading to marked reductions in caregivers' health and quality of life (QOL). Reducing CG distress has the potential to improve CG mental and physical health, improve overall QOL, and lead to improvements in the care they provide.

However, few effective interventions that can be widely delivered and easily adhered to have been rigorously evaluated. Qigong is an increasingly popular multi-modal mind-body exercise that shows promise in addressing a broad range of psychosocial and physical factors highly relevant to CGs. Sharing many characteristics with Tai Chi, Qigong incorporates elements of slow gentle movement, breath training, and number of cognitive skills including heightened body awareness, focused mental attention, and imagery-which collectively may afford greater benefits to health compared to unimodal therapies. A robust evidence base supports that Qigong and Tai Chi training in groups can improve multiple domains of physical and emotional health, QOL, and selfefficacy in diverse populations. Of note, recent national surveys indicate that a significant proportion of the US population that report using Qigong and Tai Chi for health preferred self-directed learning from DVDs and internet resources. While a handful of studies support the potential for web-based or DVD-based learning of mind-body practices, evaluations of such programs have not been well-tested, especially in CGs.

Using cancer caregivers (CCGs) as a representative population of the larger CG population, the longterm goal is to conduct a definitive trial evaluating a widely accessible and previously studied Qigong regimen (Eight Brocades, Baduanjin Qigong). Interventions will be delivered either in community-based groups led by instructors or via internet to individuals learning through recorded guided instruction supplemented with intermittent virtual live feedback from instructors. Outcomes will include QOL, fatigue, sleep disturbances, psychological distress, caregiver burden, and physical function. The short-term goals of this R34 are to conduct a mixed-methods pilot randomized controlled trial (RCT) to inform the feasibility and design of a definitive trial. The investigators will address these goals by randomizing (1:1:1) 54 CCGs to one of three conditions: (1) a community-based qigong program; (2) an internet-based qigong program; or (3) a self-care control group.

Specific Aim 1 is to finalize Qigong intervention content and delivery protocols. Specific Aim 2 will assess the 'learnability' of Qigong delivered in community-based group classes and via a web-based protocol using a novel proficiency instrument. Specific Aim 3 will evaluate the feasibility of recruiting and retaining CCGs into a 12-week clinical trial, and completing all outcomes testing protocols. Study feasibility and merit will be further informed by formal qualitative analysis of exit interviews of study completers, participants that withdraw, and Qigong instructors.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a spouse, partner, family member, or friend providing physical, emotional, and/or financial support for a cancer patient.
* Participant is able to understand, speak, and read English.
* Participant has a minimum level of 3 on the National Comprehensive Cancer Network's (NCCN) Distress Thermometer adapted for caregivers.
* Participant is able to provide informed consent.

Exclusion Criteria:

* Participant does not have an unstable illness (e.g., recent hospitalization, unstable cardiovascular disease, active cancer).
* Participant does not have a psychiatric disorders (e.g., unmanaged depression or psychosis, substance abuse, severe personality disorder)
* Participant does not have a degenerative neuromuscular condition (e.g., Parkinson's disease, multiple sclerosis).
* Participant does not have an inability to walk continuously for 15 minutes.
* Participant does not have a recent history of attending regular Qigong or similar (e.g., yoga or Tai Chi) classes defined as 20 or more classes in the past 6 months.
* Participation is not currently engaged in more than 240 minutes of moderate-intensity exercise per week.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Eligibility of recruited participants | 6 months
  Eligibility assessed by the % of eligible participants that are willing to consent to participate in the study.
Adherence to Intervention | 6 months
  Intervention adherence assessed by the rate of compliance with classes and home practice.

SECONDARY OUTCOMES:
Center for Epidemiological Studies Depression Scale Revised (CESD-R-10) | 6 months
  Self-report measure of depression consisting of 10-items. Total score is calculated based on the sum of 10 items. Each item is scored 0 to 3 yielding a total between 0 and 30. Any score equal to or greater than 10 is considered depressed.
Brief Fatigue Inventory (BFI) | 6 months
  Self-report measure of fatigue consisting of 9 items measuring the severity of fatigue and the impact of fatigue on daily functioning in the past 24 hours. Each item is scored 0-10 where 0 is no fatigue and 10 is bad fatigue, yielding a total between 0 and 90.
Pittsburgh Sleep Quality Index (PSQI), Sleep Disturbances | 6 months
  Self-report measure of sleep disturbance consisting of 19 items measuring patients' sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleeping medication use, and daytime dysfunction over the past month. Seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed up to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Caregiver Burden Scale (CBS) | 6 months
  Self-report measure of caregiver burden consisting of 22 items measuring the impact of caregiving on three dimensions of burden: objective, subjective demand, and subjective stress. Each item is scored 0-4 (0=never; 4=nearly always), yielding a total between 0 and 88. Higher scores represent a worse outcome.
Godin Leisure-Time Exercise Questionnaire, Physical Activity | 6 months
  Self-report measure of exercise consisting of 4 items measuring the frequency of light-intensity, moderate-intensity, and vigorous-intensity leisure-time physical activity. Each item is scored using units for strenuous exercise, moderate exercise, and mild exercise. Higher units represent a better outcome.
Self-Efficacy Scale, Exercise Self-Efficacy | 6 months
  Self-report measure of self-efficacy consisting of 9 items measuring self-efficacy expectations related to the ability to continue exercising in the face of barriers to exercise. Each item is scored 0-10 (0 = not confident; 10 = very confident), yielding a total between 0 and 90. Higher values represent a better outcome.
Cognitive Function, Test 1 | 6 months
  Digit Span. Participants will be asked to repeat numbers in a specific order. Performance is indicated by the average number of digits correctly remembered.
Cognitive Function, Test 2 | 6 months
  Trail Making Test Parts A & B. Participants are timed as they connect 25 circles without lifting the pen or pencil from the paper.
Physical Function, Test 1 | 6 months
  Grip strength: Strength of the dominant hand will be measured using a Jamar hydraulic hand dynamometer (Patterson Medical - Canada, Mississauga, ON, CAN).
Physical Function, Test 2 | 6 months
  Sit-to-stand. Participants will be asked to sit in a chair, cross their arms over their chest, and stand without the assistance of their arms. Number of times this is completed in 30 seconds will be recorded.
Physical Function, Test 3 | 6 months
  Balance. Participants will perform a static single-leg postural control balance test twice, once with eyes open and once with eyes closed. The maximum time for both will be limited to 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Pinky Budhrani-Shani, PhD, MSN, RN, Principal Investigator — University of Houston; Peter Wayne, PhD, Principal Investigator — Brigham and Women's Hospital and Harvard Medical School
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Alliance for Caregiving and AARP. Caregiving in the U.S. 2015. 2015; Available from: http://www.aarp.org/content/dam/aarp/ppi/2015/caregiving-in-the-united-states-2015-report-revised.pdf.
- [Background] Lambert SD, Harrison JD, Smith E, Bonevski B, Carey M, Lawsin C, Paul C, Girgis A. The unmet needs of partners and caregivers of adults diagnosed with cancer: a systematic review. BMJ Support Palliat Care. 2012 Sep;2(3):224-30. doi: 10.1136/bmjspcare-2012-000226. Epub 2012 Jul 7. PMID 24654195
- [Background] Merckaert I, Libert Y, Lieutenant F, Moucheux A, Farvacques C, Slachmuylder JL, Razavi D. Desire for formal psychological support among caregivers of patients with cancer: prevalence and implications for screening their needs. Psychooncology. 2013 Jun;22(6):1389-95. doi: 10.1002/pon.3153. Epub 2012 Aug 8. PMID 22888079
- [Background] Braun M, Mikulincer M, Rydall A, Walsh A, Rodin G. Hidden morbidity in cancer: spouse caregivers. J Clin Oncol. 2007 Oct 20;25(30):4829-34. doi: 10.1200/JCO.2006.10.0909. PMID 17947732
- [Background] Kim Y, Kashy DA, Spillers RL, Evans TV. Needs assessment of family caregivers of cancer survivors: three cohorts comparison. Psychooncology. 2010 Jun;19(6):573-82. doi: 10.1002/pon.1597. PMID 19582798
- [Background] Rabin EG, Heldt E, Hirakata VN, Bittelbrunn AC, Chachamovich E, Fleck MP. Depression and perceptions of quality of life of breast cancer survivors and their male partners. Oncol Nurs Forum. 2009 May;36(3):E153-8. doi: 10.1188/09.ONF.E153-E158. PMID 19403443
- [Background] Ploeg J, Markle-Reid M, Valaitis R, McAiney C, Duggleby W, Bartholomew A, Sherifali D. Web-Based Interventions to Improve Mental Health, General Caregiving Outcomes, and General Health for Informal Caregivers of Adults With Chronic Conditions Living in the Community: Rapid Evidence Review. J Med Internet Res. 2017 Jul 28;19(7):e263. doi: 10.2196/jmir.7564. PMID 28754652
- [Background] Lengacher CA, Reich RR, Paterson CL, Ramesar S, Park JY, Alinat C, Johnson-Mallard V, Moscoso M, Budhrani-Shani P, Miladinovic B, Jacobsen PB, Cox CE, Goodman M, Kip KE. Examination of Broad Symptom Improvement Resulting From Mindfulness-Based Stress Reduction in Breast Cancer Survivors: A Randomized Controlled Trial. J Clin Oncol. 2016 Aug 20;34(24):2827-34. doi: 10.1200/JCO.2015.65.7874. Epub 2016 May 31. PMID 27247219
- [Background] Leung L, Han H, Martin M, Kotecha J. Mindfulness-based stress reduction (MBSR) as sole intervention for non-somatisation chronic non-cancer pain (CNCP): protocol for a systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2015 May 18;5(5):e007650. doi: 10.1136/bmjopen-2015-007650. PMID 25986638
- [Background] Zeng Y, Luo T, Xie H, Huang M, Cheng AS. Health benefits of qigong or tai chi for cancer patients: a systematic review and meta-analyses. Complement Ther Med. 2014 Feb;22(1):173-86. doi: 10.1016/j.ctim.2013.11.010. Epub 2013 Dec 18. PMID 24559833
- [Background] Bajaj JS, Ellwood M, Ainger T, Burroughs T, Fagan A, Gavis EA, Heuman DM, Fuchs M, John B, Wade JB. Mindfulness-Based Stress Reduction Therapy Improves Patient and Caregiver-Reported Outcomes in Cirrhosis. Clin Transl Gastroenterol. 2017 Jul 27;8(7):e108. doi: 10.1038/ctg.2017.38. PMID 28749453
- [Background] Stjernsward S, Hansson L. Effectiveness and Usability of a Web-Based Mindfulness Intervention for Families Living with Mental Illness. Mindfulness (N Y). 2017;8(3):751-764. doi: 10.1007/s12671-016-0653-2. Epub 2016 Dec 8. PMID 28515801
- [Background] Milbury K, Chaoul A, Engle R, Liao Z, Yang C, Carmack C, Shannon V, Spelman A, Wangyal T, Cohen L. Couple-based Tibetan yoga program for lung cancer patients and their caregivers. Psychooncology. 2015 Jan;24(1):117-20. doi: 10.1002/pon.3588. Epub 2014 May 29. No abstract available. PMID 24890852
- [Background] Milbury K, Mallaiah S, Mahajan A, Armstrong T, Weathers SP, Moss KE, Goktepe N, Spelman A, Cohen L. Yoga Program for High-Grade Glioma Patients Undergoing Radiotherapy and Their Family Caregivers. Integr Cancer Ther. 2018 Jun;17(2):332-336. doi: 10.1177/1534735417689882. Epub 2017 Feb 2. PMID 28150503
- [Background] Kotronoulas G, Wengstrom Y, Kearney N. Alterations and Interdependence in Self-Reported Sleep-Wake Parameters of Patient-Caregiver Dyads During Adjuvant Chemotherapy for Breast Cancer . Oncol Nurs Forum. 2016 May 1;43(3):288-301. doi: 10.1188/16.ONF.288-301. PMID 27105191
- [Background] von Heymann-Horan AB, Puggaard LB, Nissen KG, Benthien KS, Bidstrup P, Coyne J, Johansen C, Kjellberg J, Nordly M, Sjogren P, Timm H, von der Maase H, Guldin MB. Dyadic psychological intervention for patients with cancer and caregivers in home-based specialized palliative care: The Domus model. Palliat Support Care. 2018 Apr;16(2):189-197. doi: 10.1017/S1478951517000141. Epub 2017 Mar 30. PMID 28357972
- [Background] Whitebird RR, Kreitzer M, Crain AL, Lewis BA, Hanson LR, Enstad CJ. Mindfulness-based stress reduction for family caregivers: a randomized controlled trial. Gerontologist. 2013 Aug;53(4):676-86. doi: 10.1093/geront/gns126. Epub 2012 Oct 15. PMID 23070934
- [Background] Wayne P. M., and Fuerst. M. The Harvard Medical School Guide to Tai Chi: 12 Weeks to a Healthy Body, Strong Heart & Sharp Mind. 2013, Boston: Shambhala Publications Inc.
- [Background] Wayne PM, Berkowitz DL, Litrownik DE, Buring JE, Yeh GY. What do we really know about the safety of tai chi?: A systematic review of adverse event reports in randomized trials. Arch Phys Med Rehabil. 2014 Dec;95(12):2470-83. doi: 10.1016/j.apmr.2014.05.005. Epub 2014 May 27. PMID 24878398
- [Background] Wayne PM, Hausdorff JM, Lough M, Gow BJ, Lipsitz L, Novak V, Macklin EA, Peng CK, Manor B. Tai Chi Training may Reduce Dual Task Gait Variability, a Potential Mediator of Fall Risk, in Healthy Older Adults: Cross-Sectional and Randomized Trial Studies. Front Hum Neurosci. 2015 Jun 9;9:332. doi: 10.3389/fnhum.2015.00332. eCollection 2015. PMID 26106316
- [Background] Song R, Grabowska W, Park M, Osypiuk K, Vergara-Diaz GP, Bonato P, Hausdorff JM, Fox M, Sudarsky LR, Macklin E, Wayne PM. The impact of Tai Chi and Qigong mind-body exercises on motor and non-motor function and quality of life in Parkinson's disease: A systematic review and meta-analysis. Parkinsonism Relat Disord. 2017 Aug;41:3-13. doi: 10.1016/j.parkreldis.2017.05.019. Epub 2017 May 25. PMID 28602515
- [Background] Zou L, SasaKi JE, Wang H, Xiao Z, Fang Q, Zhang M. A Systematic Review and Meta-Analysis Baduanjin Qigong for Health Benefits: Randomized Controlled Trials. Evid Based Complement Alternat Med. 2017;2017:4548706. doi: 10.1155/2017/4548706. Epub 2017 Mar 7. PMID 28367223
- [Background] Budhrani-Shani P, Berry DL, Arcari P, Langevin H, Wayne PM. Mind-Body Exercises for Nurses with Chronic Low Back Pain: An Evidence-Based Review. Nurs Res Pract. 2016;2016:9018036. doi: 10.1155/2016/9018036. Epub 2016 Jul 3. PMID 27446610
- [Background] Lauche R, Wayne PM, Dobos G, Cramer H. Prevalence, Patterns, and Predictors of T'ai Chi and Qigong Use in the United States: Results of a Nationally Representative Survey. J Altern Complement Med. 2016 Apr;22(4):336-42. doi: 10.1089/acm.2015.0356. Epub 2016 Mar 16. PMID 26981616
- [Background] Chen HH, Yeh ML, Lee FY. The effects of Baduanjin qigong in the prevention of bone loss for middle-aged women. Am J Chin Med. 2006;34(5):741-7. doi: 10.1142/S0192415X06004259. PMID 17080541
- [Background] Tao J, Chen X, Egorova N, Liu J, Xue X, Wang Q, Zheng G, Li M, Hong W, Sun S, Chen L, Kong J. Tai Chi Chuan and Baduanjin practice modulates functional connectivity of the cognitive control network in older adults. Sci Rep. 2017 Feb 7;7:41581. doi: 10.1038/srep41581. PMID 28169310
- [Background] Bevans M, Sternberg EM. Caregiving burden, stress, and health effects among family caregivers of adult cancer patients. JAMA. 2012 Jan 25;307(4):398-403. doi: 10.1001/jama.2012.29. PMID 22274687
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Hiseman JP, Fackrell R. Caregiver Burden and the Nonmotor Symptoms of Parkinson's Disease. Int Rev Neurobiol. 2017;133:479-497. doi: 10.1016/bs.irn.2017.05.035. Epub 2017 Jul 21. PMID 28802929
- [Background] Schulz R, Beach SR. Caregiving as a risk factor for mortality: the Caregiver Health Effects Study. JAMA. 1999 Dec 15;282(23):2215-9. doi: 10.1001/jama.282.23.2215. PMID 10605972
- [Background] Haines J, Spadaro KC, Choi J, Hoffman LA, Blazeck AM. Reducing stress and anxiety in caregivers of lung transplant patients: benefits of mindfulness meditation. Int J Organ Transplant Med. 2014;5(2):50-6. PMID 25013679
- [Background] Caqueo-Urizar A, Alessandrini M, Urzua A, Zendjidjian X, Boyer L, Williams DR. Caregiver's quality of life and its positive impact on symptomatology and quality of life of patients with schizophrenia. Health Qual Life Outcomes. 2017 Apr 19;15(1):76. doi: 10.1186/s12955-017-0652-6. PMID 28424076
- [Background] Bluethmann SM, Mariotto AB, Rowland JH. Anticipating the "Silver Tsunami": Prevalence Trajectories and Comorbidity Burden among Older Cancer Survivors in the United States. Cancer Epidemiol Biomarkers Prev. 2016 Jul;25(7):1029-36. doi: 10.1158/1055-9965.EPI-16-0133. PMID 27371756
- [Background] Given BA, Given CW, Sherwood P. The challenge of quality cancer care for family caregivers. Semin Oncol Nurs. 2012 Nov;28(4):205-12. doi: 10.1016/j.soncn.2012.09.002. PMID 23107177
- [Background] Romito F, Goldzweig G, Cormio C, Hagedoorn M, Andersen BL. Informal caregiving for cancer patients. Cancer. 2013 Jun 1;119 Suppl 11(0 11):2160-9. doi: 10.1002/cncr.28057. PMID 23695928
- [Background] Kim Y, Shaffer KM, Carver CS, Cannady RS. Quality of life of family caregivers 8 years after a relative's cancer diagnosis: follow-up of the National Quality of Life Survey for Caregivers. Psychooncology. 2016 Mar;25(3):266-74. doi: 10.1002/pon.3843. Epub 2015 May 15. PMID 25976620
- [Background] Copley Cobb S, Etkins L, Nelson M, Egleston B, Sweeney CW. A Comparison of the Reactions of Caregivers of Patients With Cancer Versus Patients With Other Chronic Medical Conditions. Oncol Nurs Forum. 2016 May 1;43(3):321-7. doi: 10.1188/16.ONF.321-327. PMID 27105193
- [Background] Shaffer KM, Kim Y, Carver CS, Cannady RS. Effects of caregiving status and changes in depressive symptoms on development of physical morbidity among long-term cancer caregivers. Health Psychol. 2017 Aug;36(8):770-778. doi: 10.1037/hea0000528. Epub 2017 Jun 22. PMID 28639819
- [Background] Williams AL. Family Caregivers to Adults with Cancer: The Consequences of Caring. Recent Results Cancer Res. 2018;210:87-103. doi: 10.1007/978-3-319-64310-6_6. PMID 28924681
- [Background] Zarit SH. Behavioral disturbances of dementia and caregiver issues. Int Psychogeriatr. 1996;8 Suppl 3:263-8; discussion 269-72. doi: 10.1017/s1041610297003451. No abstract available. PMID 9154574
- [Background] Northouse LL, Katapodi MC, Song L, Zhang L, Mood DW. Interventions with family caregivers of cancer patients: meta-analysis of randomized trials. CA Cancer J Clin. 2010 Sep-Oct;60(5):317-39. doi: 10.3322/caac.20081. Epub 2010 Aug 13. PMID 20709946
- [Background] Northouse LL, Katapodi MC, Schafenacker AM, Weiss D. The impact of caregiving on the psychological well-being of family caregivers and cancer patients. Semin Oncol Nurs. 2012 Nov;28(4):236-45. doi: 10.1016/j.soncn.2012.09.006. PMID 23107181
- [Background] Lin CR, Chen SC, Chang JT, Fang YY, Lai YH. Fear of Cancer Recurrence and Its Impacts on Quality of Life in Family Caregivers of Patients With Head and Neck Cancers. J Nurs Res. 2016 Sep;24(3):240-8. doi: 10.1097/jnr.0000000000000169. PMID 27509212
- [Background] Maguire R, Hanly P, Balfe M, Timmons A, Hyland P, O'Sullivan E, Butow P, Sharp L. Worry in Head and Neck Cancer Caregivers: The Role of Survivor Factors, Care-Related Stressors, and Loneliness in Predicting Fear of Recurrence. Nurs Res. 2017 Jul/Aug;66(4):295-303. doi: 10.1097/NNR.0000000000000223. PMID 28654567
- [Background] Lee S, Colditz GA, Berkman LF, Kawachi I. Caregiving and risk of coronary heart disease in U.S. women: a prospective study. Am J Prev Med. 2003 Feb;24(2):113-9. doi: 10.1016/s0749-3797(02)00582-2. PMID 12568816
- [Background] Gouin JP, Hantsoo L, Kiecolt-Glaser JK. Immune dysregulation and chronic stress among older adults: a review. Neuroimmunomodulation. 2008;15(4-6):251-9. doi: 10.1159/000156468. Epub 2008 Nov 26. PMID 19047802
- [Background] Suzuki K, Tamakoshi K, Sakakibara H. Caregiving activities closely associated with the development of low-back pain among female family caregivers. J Clin Nurs. 2016 Aug;25(15-16):2156-67. doi: 10.1111/jocn.13167. Epub 2016 Apr 22. PMID 27105394
- [Background] Sharan D, Ajeesh PS, Rameshkumar R, Manjula M. Musculoskeletal disorders in caregivers of children with cerebral palsy following a multilevel surgery. Work. 2012;41 Suppl 1:1891-5. doi: 10.3233/WOR-2012-0403-1891. PMID 22316991
- [Background] Cho HJ, Lavretsky H, Olmstead R, Levin MJ, Oxman MN, Irwin MR. Sleep disturbance and depression recurrence in community-dwelling older adults: a prospective study. Am J Psychiatry. 2008 Dec;165(12):1543-50. doi: 10.1176/appi.ajp.2008.07121882. Epub 2008 Sep 2. PMID 18765482
- [Background] Wayne P. M., F.M.L., The Harvard Medical School Guide to Tai Chi: 12 Weeks to a healthy body, strong heart, and sharp mind. . 2012, Boston, MA: Harvard Health Publications.
- [Background] Dharmawardene M, Givens J, Wachholtz A, Makowski S, Tjia J. A systematic review and meta-analysis of meditative interventions for informal caregivers and health professionals. BMJ Support Palliat Care. 2016 Jun;6(2):160-9. doi: 10.1136/bmjspcare-2014-000819. Epub 2015 Mar 26. PMID 25812579
- [Background] Lavretsky H, Epel ES, Siddarth P, Nazarian N, Cyr NS, Khalsa DS, Lin J, Blackburn E, Irwin MR. A pilot study of yogic meditation for family dementia caregivers with depressive symptoms: effects on mental health, cognition, and telomerase activity. Int J Geriatr Psychiatry. 2013 Jan;28(1):57-65. doi: 10.1002/gps.3790. Epub 2012 Mar 11. PMID 22407663
- [Background] Lavretsky H, Siddarth P, Irwin MR. Improving depression and enhancing resilience in family dementia caregivers: a pilot randomized placebo-controlled trial of escitalopram. Am J Geriatr Psychiatry. 2010 Feb;18(2):154-62. doi: 10.1097/JGP.0b013e3181beab1e. PMID 20104071
- [Background] Carlson LE, Zelinski E, Toivonen K, Flynn M, Qureshi M, Piedalue KA, Grant R. Mind-Body Therapies in Cancer: What Is the Latest Evidence? Curr Oncol Rep. 2017 Aug 18;19(10):67. doi: 10.1007/s11912-017-0626-1. PMID 28822063
- [Background] Cheng FK. Effects of Baduanjin on mental health: a comprehensive review. J Bodyw Mov Ther. 2015 Jan;19(1):138-49. doi: 10.1016/j.jbmt.2014.11.001. Epub 2014 Nov 11. PMID 25603754
- [Background] Chan JS, Ho RT, Chung KF, Wang CW, Yao TJ, Ng SM, Chan CL. Qigong exercise alleviates fatigue, anxiety, and depressive symptoms, improves sleep quality, and shortens sleep latency in persons with chronic fatigue syndrome-like illness. Evid Based Complement Alternat Med. 2014;2014:106048. doi: 10.1155/2014/106048. Epub 2014 Dec 25. PMID 25610473
- [Background] Jiang YH, Tan C, Yuan S. RETRACTED ARTICLE: Baduanjin Exercise for Insomnia: A Systematic Review and Meta-Analysis. Behav Sleep Med. 2023 May-Jun;21(3):i-xiii. doi: 10.1080/15402002.2017.1363042. Epub 2017 Sep 15. PMID 28777659
- [Background] Li M, Fang Q, Li J, Zheng X, Tao J, Yan X, Lin Q, Lan X, Chen B, Zheng G, Chen L. The Effect of Chinese Traditional Exercise-Baduanjin on Physical and Psychological Well-Being of College Students: A Randomized Controlled Trial. PLoS One. 2015 Jul 9;10(7):e0130544. doi: 10.1371/journal.pone.0130544. eCollection 2015. PMID 26158769
- [Background] Bai Z, Guan Z, Fan Y, Liu C, Yang K, Ma B, Wu B. The Effects of Qigong for Adults with Chronic Pain: Systematic Review and Meta-Analysis. Am J Chin Med. 2015;43(8):1525-39. doi: 10.1142/S0192415X15500871. Epub 2015 Nov 30. PMID 26621441
- [Background] Lauche R, Cramer H, Hauser W, Dobos G, Langhorst J. A systematic review and meta-analysis of qigong for the fibromyalgia syndrome. Evid Based Complement Alternat Med. 2013;2013:635182. doi: 10.1155/2013/635182. Epub 2013 Oct 31. PMID 24288564
- [Background] Lee MS, Pittler MH, Ernst E. External qigong for pain conditions: a systematic review of randomized clinical trials. J Pain. 2007 Nov;8(11):827-31. doi: 10.1016/j.jpain.2007.05.016. Epub 2007 Aug 9. PMID 17690012
- [Background] Lee MS, Pittler MH, Ernst E. Internal qigong for pain conditions: a systematic review. J Pain. 2009 Nov;10(11):1121-1127.e14. doi: 10.1016/j.jpain.2009.03.009. Epub 2009 Jun 25. PMID 19559656
- [Background] Buric I, Farias M, Jong J, Mee C, Brazil IA. What Is the Molecular Signature of Mind-Body Interventions? A Systematic Review of Gene Expression Changes Induced by Meditation and Related Practices. Front Immunol. 2017 Jun 16;8:670. doi: 10.3389/fimmu.2017.00670. eCollection 2017. PMID 28670311
- [Background] Oh B, Butow PN, Mullan BA, Clarke SJ, Beale PJ, Pavlakis N, Lee MS, Rosenthal DS, Larkey L, Vardy J. Effect of medical Qigong on cognitive function, quality of life, and a biomarker of inflammation in cancer patients: a randomized controlled trial. Support Care Cancer. 2012 Jun;20(6):1235-42. doi: 10.1007/s00520-011-1209-6. Epub 2011 Jun 19. PMID 21688163
- [Background] Chen MC, Liu HE, Huang HY, Chiou AF. The effect of a simple traditional exercise programme (Baduanjin exercise) on sleep quality of older adults: a randomized controlled trial. Int J Nurs Stud. 2012 Mar;49(3):265-73. doi: 10.1016/j.ijnurstu.2011.09.009. Epub 2011 Sep 29. PMID 21963235
- [Background] Ho RTH, Wan AHY, Chan JSM, Ng SM, Chung KF, Chan CLW. Study protocol on comparative effectiveness of mindfulness meditation and qigong on psychophysiological outcomes for patients with colorectal cancer: a randomized controlled trial. BMC Complement Altern Med. 2017 Aug 8;17(1):390. doi: 10.1186/s12906-017-1898-6. PMID 28789681
- [Background] Xiao CM, Zhuang YC. Effect of health Baduanjin Qigong for mild to moderate Parkinson's disease. Geriatr Gerontol Int. 2016 Aug;16(8):911-9. doi: 10.1111/ggi.12571. Epub 2015 Aug 26. PMID 26310941
- [Background] Kushner RF, Sorensen KW. Lifestyle medicine: the future of chronic disease management. Curr Opin Endocrinol Diabetes Obes. 2013 Oct;20(5):389-95. doi: 10.1097/01.med.0000433056.76699.5d. PMID 23974765
- [Background] Katrancha ED, Hoffman LA, Zullo TG, Tuite PK, Garand L. Effects of a video guided T'ai Chi group intervention on center of balance and falls efficacy: a pilot study. Geriatr Nurs. 2015 Jan-Feb;36(1):9-14. doi: 10.1016/j.gerinurse.2014.08.015. PMID 25660190
- [Background] Dam AEH, van Boxtel MPJ, Rozendaal N, Verhey FRJ, de Vugt ME. Development and feasibility of Inlife: A pilot study of an online social support intervention for informal caregivers of people with dementia. PLoS One. 2017 Sep 8;12(9):e0183386. doi: 10.1371/journal.pone.0183386. eCollection 2017. PMID 28886056
- [Background] Wu G, Keyes LM. Group tele-exercise for improving balance in elders. Telemed J E Health. 2006 Oct;12(5):561-70. doi: 10.1089/tmj.2006.12.561. PMID 17042710
- [Background] Wu G, Keyes L, Callas P, Ren X, Bookchin B. Comparison of telecommunication, community, and home-based Tai Chi exercise programs on compliance and effectiveness in elders at risk for falls. Arch Phys Med Rehabil. 2010 Jun;91(6):849-56. doi: 10.1016/j.apmr.2010.01.024. PMID 20510973
- [Background] Sannes TS, Mansky PJ, Chesney MA. The need for attention to dose in mind-body interventions: lessons from t'ai chi clinical trials. J Altern Complement Med. 2008 Jul;14(6):645-53. doi: 10.1089/acm.2007.0680. PMID 18684072
- [Background] Wayne PM, Kaptchuk TJ. Challenges inherent to t'ai chi research: part I--t'ai chi as a complex multicomponent intervention. J Altern Complement Med. 2008 Jan-Feb;14(1):95-102. doi: 10.1089/acm.2007.7170a. PMID 18199021
- [Background] Wayne PM, Kaptchuk TJ. Challenges inherent to t'ai chi research: part II-defining the intervention and optimal study design. J Altern Complement Med. 2008 Mar;14(2):191-7. doi: 10.1089/acm.2007.7170b. PMID 18446928
- [Background] Moy ML, Wayne PM, Litrownik D, Beach D, Klings ES, Davis RB, Yeh GY. Long-term Exercise After Pulmonary Rehabilitation (LEAP): Design and rationale of a randomized controlled trial of Tai Chi. Contemp Clin Trials. 2015 Nov;45(Pt B):458-467. doi: 10.1016/j.cct.2015.09.004. Epub 2015 Sep 8. PMID 26362690
- [Background] Salmoirago-Blotcher E, Wayne P, Bock BC, Dunsiger S, Wu WC, Stabile L, Yeh G. Design and methods of the Gentle Cardiac Rehabilitation Study--A behavioral study of tai chi exercise for patients not attending cardiac rehabilitation. Contemp Clin Trials. 2015 Jul;43:243-51. doi: 10.1016/j.cct.2015.06.020. Epub 2015 Jun 24. PMID 26115880
- [Background] Salmoirago-Blotcher E, Wayne PM, Dunsiger S, Krol J, Breault C, Bock BC, Wu WC, Yeh GY. Tai Chi Is a Promising Exercise Option for Patients With Coronary Heart Disease Declining Cardiac Rehabilitation. J Am Heart Assoc. 2017 Oct 11;6(10):e006603. doi: 10.1161/JAHA.117.006603. PMID 29021268
- [Background] Wayne PM, Gow BJ, Costa MD, Peng CK, Lipsitz LA, Hausdorff JM, Davis RB, Walsh JN, Lough M, Novak V, Yeh GY, Ahn AC, Macklin EA, Manor B. Complexity-Based Measures Inform Effects of Tai Chi Training on Standing Postural Control: Cross-Sectional and Randomized Trial Studies. PLoS One. 2014 Dec 10;9(12):e114731. doi: 10.1371/journal.pone.0114731. eCollection 2014. PMID 25494333
- [Background] Yeh GY, Chan CW, Wayne PM, Conboy L. The Impact of Tai Chi Exercise on Self-Efficacy, Social Support, and Empowerment in Heart Failure: Insights from a Qualitative Sub-Study from a Randomized Controlled Trial. PLoS One. 2016 May 13;11(5):e0154678. doi: 10.1371/journal.pone.0154678. eCollection 2016. PMID 27177041
- [Background] Yeh GY, Mu L, Davis RB, Wayne PM. Correlates of Exercise Self-efficacy in a Randomized Trial of Mind-Body Exercise in Patients With Chronic Heart Failure. J Cardiopulm Rehabil Prev. 2016 May-Jun;36(3):186-94. doi: 10.1097/HCR.0000000000000170. PMID 26959498
- [Background] Yeh GY, Wayne PM, Litrownik D, Roberts DH, Davis RB, Moy ML. Tai chi mind-body exercise in patients with COPD: study protocol for a randomized controlled trial. Trials. 2014 Aug 28;15:337. doi: 10.1186/1745-6215-15-337. PMID 25168853
- [Background] Yeung AS, Feng R, Kim DJH, Wayne PM, Yeh GY, Baer L, Lee OE, Denninger JW, Benson H, Fricchione GL, Alpert J, Fava M. A Pilot, Randomized Controlled Study of Tai Chi With Passive and Active Controls in the Treatment of Depressed Chinese Americans. J Clin Psychiatry. 2017 May;78(5):e522-e528. doi: 10.4088/JCP.16m10772. PMID 28570792
- [Background] Budhrani PH, Lengacher CA, Kip K, Tofthagen C, Jim H. An integrative review of subjective and objective measures of sleep disturbances in breast cancer survivors. Clin J Oncol Nurs. 2015 Apr;19(2):185-91. doi: 10.1188/15.CJON.185-191. PMID 25840384
- [Background] Budhrani PH, Lengacher CA, Kip KE, Tofthagen C, Jim H. Minority Breast Cancer Survivors: The Association between Race/Ethnicity, Objective Sleep Disturbances, and Physical and Psychological Symptoms. Nurs Res Pract. 2014;2014:858403. doi: 10.1155/2014/858403. Epub 2014 Jul 2. PMID 25101174
- [Background] Lengacher CA, Johnson-Mallard V, Barta M, Fitzgerald S, Moscoso MS, Post-White J, Jacobsen PB, Molinari Shelton M, Le N, Budhrani P, Goodman M, Kip KE. Feasibility of a mindfulness-based stress reduction program for early-stage breast cancer survivors. J Holist Nurs. 2011 Jun;29(2):107-17. doi: 10.1177/0898010110385938. Epub 2010 Nov 1. PMID 21041554
- [Background] Lengacher CA, Reich RR, Kip KE, Barta M, Ramesar S, Paterson CL, Moscoso MS, Carranza I, Budhrani PH, Kim SJ, Park HY, Jacobsen PB, Schell MJ, Jim HS, Post-White J, Farias JR, Park JY. Influence of mindfulness-based stress reduction (MBSR) on telomerase activity in women with breast cancer (BC). Biol Res Nurs. 2014 Oct;16(4):438-47. doi: 10.1177/1099800413519495. Epub 2014 Jan 30. PMID 24486564
- [Background] Lengacher CA, Reich RR, Paterson CL, Jim HS, Ramesar S, Alinat CB, Budhrani PH, Farias JR, Shelton MM, Moscoso MS, Park JY, Kip KE. The effects of mindfulness-based stress reduction on objective and subjective sleep parameters in women with breast cancer: a randomized controlled trial. Psychooncology. 2015 Apr;24(4):424-32. doi: 10.1002/pon.3603. Epub 2014 Jun 18. PMID 24943918
- [Background] Lengacher CA, Reich RR, Post-White J, Moscoso M, Shelton MM, Barta M, Le N, Budhrani P. Mindfulness based stress reduction in post-treatment breast cancer patients: an examination of symptoms and symptom clusters. J Behav Med. 2012 Feb;35(1):86-94. doi: 10.1007/s10865-011-9346-4. Epub 2011 Apr 20. PMID 21506018
- [Background] Lengacher CA, Shelton MM, Reich RR, Barta MK, Johnson-Mallard V, Moscoso MS, Paterson C, Ramesar S, Budhrani P, Carranza I, Lucas J, Jacobsen PB, Goodman MJ, Kip KE. Mindfulness based stress reduction (MBSR(BC)) in breast cancer: evaluating fear of recurrence (FOR) as a mediator of psychological and physical symptoms in a randomized control trial (RCT). J Behav Med. 2014 Apr;37(2):185-95. doi: 10.1007/s10865-012-9473-6. Epub 2012 Nov 27. PMID 23184061
- [Background] McQuade JL, Prinsloo S, Chang DZ, Spelman A, Wei Q, Basen-Engquist K, Harrison C, Zhang Z, Kuban D, Lee A, Cohen L. Qigong/tai chi for sleep and fatigue in prostate cancer patients undergoing radiotherapy: a randomized controlled trial. Psychooncology. 2017 Nov;26(11):1936-1943. doi: 10.1002/pon.4256. Epub 2016 Sep 20. PMID 27548839
- [Background] Yeh GY, Wood MJ, Lorell BH, Stevenson LW, Eisenberg DM, Wayne PM, Goldberger AL, Davis RB, Phillips RS. Effects of tai chi mind-body movement therapy on functional status and exercise capacity in patients with chronic heart failure: a randomized controlled trial. Am J Med. 2004 Oct 15;117(8):541-8. doi: 10.1016/j.amjmed.2004.04.016. PMID 15465501
- [Background] Yeh GY, McCarthy EP, Wayne PM, Stevenson LW, Wood MJ, Forman D, Davis RB, Phillips RS. Tai chi exercise in patients with chronic heart failure: a randomized clinical trial. Arch Intern Med. 2011 Apr 25;171(8):750-7. doi: 10.1001/archinternmed.2011.150. PMID 21518942
- [Background] Yeh GY, Wood MJ, Wayne PM, Quilty MT, Stevenson LW, Davis RB, Phillips RS, Forman DE. Tai chi in patients with heart failure with preserved ejection fraction. Congest Heart Fail. 2013 Mar-Apr;19(2):77-84. doi: 10.1111/chf.12005. Epub 2012 Oct 12. PMID 23057654
- [Background] Li L, Manor B. Long term Tai Chi exercise improves physical performance among people with peripheral neuropathy. Am J Chin Med. 2010;38(3):449-59. doi: 10.1142/S0192415X1000797X. PMID 20503464
- [Background] Manor B, Lipsitz LA, Wayne PM, Peng CK, Li L. Complexity-based measures inform Tai Chi's impact on standing postural control in older adults with peripheral neuropathy. BMC Complement Altern Med. 2013 Apr 16;13:87. doi: 10.1186/1472-6882-13-87. PMID 23587193
- [Background] McGibbon CA, Krebs DE, Wolf SL, Wayne PM, Scarborough DM, Parker SW. Tai Chi and vestibular rehabilitation effects on gaze and whole-body stability. J Vestib Res. 2004;14(6):467-78. PMID 15735329
- [Background] McGibbon CA, Krebs DE, Parker SW, Scarborough DM, Wayne PM, Wolf SL. Tai Chi and vestibular rehabilitation improve vestibulopathic gait via different neuromuscular mechanisms: preliminary report. BMC Neurol. 2005 Feb 18;5(1):3. doi: 10.1186/1471-2377-5-3. PMID 15717934
- [Background] Wayne PM, Manor B, Novak V, Costa MD, Hausdorff JM, Goldberger AL, Ahn AC, Yeh GY, Peng CK, Lough M, Davis RB, Quilty MT, Lipsitz LA. A systems biology approach to studying Tai Chi, physiological complexity and healthy aging: design and rationale of a pragmatic randomized controlled trial. Contemp Clin Trials. 2013 Jan;34(1):21-34. doi: 10.1016/j.cct.2012.09.006. Epub 2012 Sep 29. PMID 23026349
- [Background] Wayne PM, Kiel DP, Buring JE, Connors EM, Bonato P, Yeh GY, Cohen CJ, Mancinelli C, Davis RB. Impact of Tai Chi exercise on multiple fracture-related risk factors in post-menopausal osteopenic women: a pilot pragmatic, randomized trial. BMC Complement Altern Med. 2012 Jan 30;12:7. doi: 10.1186/1472-6882-12-7. PMID 22289280
- [Background] Yeung A, Lepoutre V, Wayne P, Yeh G, Slipp LE, Fava M, Denninger JW, Benson H, Fricchione GL. Tai chi treatment for depression in Chinese Americans: a pilot study. Am J Phys Med Rehabil. 2012 Oct;91(10):863-70. doi: 10.1097/PHM.0b013e31825f1a67. PMID 22790795
- [Background] Wayne PM, Gagnon MM, Macklin EA, Travison TG, Manor B, Lachman M, Thomas CP, Lipsitz LA. The Mind Body-Wellness in Supportive Housing (Mi-WiSH) study: Design and rationale of a cluster randomized controlled trial of Tai Chi in senior housing. Contemp Clin Trials. 2017 Sep;60:96-104. doi: 10.1016/j.cct.2017.07.005. Epub 2017 Jul 8. PMID 28694204
- [Background] Carlson LE, Zelinski EL, Speca M, Balneaves LG, Jones JM, Santa Mina D, Wayne PM, Campbell TS, Giese-Davis J, Faris P, Zwicker J, Patel K, Beattie TL, Cole S, Toivonen K, Nation J, Peng P, Thong B, Wong R, Vohra S. Protocol for the MATCH study (Mindfulness and Tai Chi for cancer health): A preference-based multi-site randomized comparative effectiveness trial (CET) of Mindfulness-Based Cancer Recovery (MBCR) vs. Tai Chi/Qigong (TCQ) for cancer survivors. Contemp Clin Trials. 2017 Aug;59:64-76. doi: 10.1016/j.cct.2017.05.015. Epub 2017 May 30. PMID 28576734
- [Background] Lengacher CA, Kip KE, Barta M, Post-White J, Jacobsen PB, Groer M, Lehman B, Moscoso MS, Kadel R, Le N, Loftus L, Stevens CA, Malafa MP, Shelton MM. A pilot study evaluating the effect of mindfulness-based stress reduction on psychological status, physical status, salivary cortisol, and interleukin-6 among advanced-stage cancer patients and their caregivers. J Holist Nurs. 2012 Sep;30(3):170-85. doi: 10.1177/0898010111435949. Epub 2012 Mar 21. PMID 22442202
- [Background] Reich RR, Lengacher CA, Alinat CB, Kip KE, Paterson C, Ramesar S, Han HS, Ismail-Khan R, Johnson-Mallard V, Moscoso M, Budhrani-Shani P, Shivers S, Cox CE, Goodman M, Park J. Mindfulness-Based Stress Reduction in Post-treatment Breast Cancer Patients: Immediate and Sustained Effects Across Multiple Symptom Clusters. J Pain Symptom Manage. 2017 Jan;53(1):85-95. doi: 10.1016/j.jpainsymman.2016.08.005. Epub 2016 Oct 5. PMID 27720794
- [Background] Rosengren KS, Christou E, Yang Y, Kass D, Boule A. Quantification of taiji learning in older adults. J Am Geriatr Soc. 2003 Aug;51(8):1186-7. doi: 10.1046/j.1532-5415.2003.51376.x. No abstract available. PMID 12890093
- [Background] Fischer M, Fugate-Woods N, Wayne PM. Use of pragmatic community-based interventions to enhance recruitment and adherence in a randomized trial of Tai Chi for women with osteopenia: insights from a qualitative substudy. Menopause. 2014 Nov;21(11):1181-9. doi: 10.1097/GME.0000000000000257. PMID 24845395
- [Background] Yeh GY, Roberts DH, Wayne PM, Davis RB, Quilty MT, Phillips RS. Tai chi exercise for patients with chronic obstructive pulmonary disease: a pilot study. Respir Care. 2010 Nov;55(11):1475-82. PMID 20979675
- [Background] Budhrani-Shani P, Chau NG, Berry DL. Psychosocial distress and the preferred method of delivery of mind-body interventions among patients with head-and-neck cancer. Patient Relat Outcome Meas. 2018 Apr 3;9:129-136. doi: 10.2147/PROM.S149978. eCollection 2018. PMID 29662331
- [Background] Wayne PM, Buring JE, Davis RB, Connors EM, Bonato P, Patritti B, Fischer M, Yeh GY, Cohen CJ, Carroll D, Kiel DP. Tai Chi for osteopenic women: design and rationale of a pragmatic randomized controlled trial. BMC Musculoskelet Disord. 2010 Mar 1;11:40. doi: 10.1186/1471-2474-11-40. PMID 20193083
- [Background] Lee, J., H. Chung-Hung, and L. Ting-Yang, A Kinect-based Tai Chi exercises evaluation system for physical rehabilitation. IEEE International Conference. 2014, Consumer Electronics.
- [Background] Kitsunezaki, N.e.a., Kinect applications for the physical rehabilitation, in IEEE International Symposium on. IEEE. 2013, Measurements and Applications Proceedings (MeMeA).
- [Background] Sasaki, A.e.a., Instruction Display for Learning Taijiquan Motions, in IEEE International Symposium on. IEEE. 2007, Industrial Electronics.
- [Background] Chua, P.T., Training for physical tasks in virtual environments: Tai Chi, in IEEE International Symposium on IEEE. 2003, Virtual Reality.
- [Background] De Morais, W. Ourique, and N. Wickstrom, A serious computer game to assist Tai Chi training for the elderly, in IEEE 1st International Conference. 2011, Serious Games and Application for Health.
- [Background] Chang JY, Tsai PF, Beck C, Hagen JL, Huff DC, Anand KJ, Roberson PK, Rosengren KS, Beuscher L. The effect of tai chi on cognition in elders with cognitive impairment. Medsurg Nurs. 2011 Mar-Apr;20(2):63-9; quiz 70. PMID 21560956
- [Background] Tsai PF, Chang JY, Beck C, Hagen J, Anand KJ, Kuo YF, Roberson PK, Rosengren K, Beuscher L. The Feasibility of Implementing Tai Chi for Nursing Home Residents With Knee Osteoarthritis and Cognitive Impairment. Act Dir Q Alzheimers Other Dement Patients. 2009 Winter;10(1):9-17. PMID 25249819
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Radloff, L., The CES-D scale: a self-report depression scale for research in the general population. Applied Psychological Measurement 1977. 1: p. 385-401.
- [Background] Mendoza TR, Wang XS, Cleeland CS, Morrissey M, Johnson BA, Wendt JK, Huber SL. The rapid assessment of fatigue severity in cancer patients: use of the Brief Fatigue Inventory. Cancer. 1999 Mar 1;85(5):1186-96. doi: 10.1002/(sici)1097-0142(19990301)85:53.0.co;2-n. PMID 10091805
- [Background] Northouse LL. Mastectomy patients and the fear of cancer recurrence. Cancer Nurs. 1981 Jun;4(3):213-20. No abstract available. PMID 6909039
- [Background] Thewes B, Butow P, Zachariae R, Christensen S, Simard S, Gotay C. Fear of cancer recurrence: a systematic literature review of self-report measures. Psychooncology. 2012 Jun;21(6):571-87. doi: 10.1002/pon.2070. Epub 2011 Oct 21. PMID 22021099
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Elmstahl S, Malmberg B, Annerstedt L. Caregiver's burden of patients 3 years after stroke assessed by a novel caregiver burden scale. Arch Phys Med Rehabil. 1996 Feb;77(2):177-82. doi: 10.1016/s0003-9993(96)90164-1. PMID 8607743
- [Background] Godin G, Belanger-Gravel A, Amireault S, Vohl MC, Perusse L. The effect of mere-measurement of cognitions on physical activity behavior: a randomized controlled trial among overweight and obese individuals. Int J Behav Nutr Phys Act. 2011 Jan 11;8:2. doi: 10.1186/1479-5868-8-2. PMID 21223565
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Kuh D, Bassey EJ, Butterworth S, Hardy R, Wadsworth ME; Musculoskeletal Study Team. Grip strength, postural control, and functional leg power in a representative cohort of British men and women: associations with physical activity, health status, and socioeconomic conditions. J Gerontol A Biol Sci Med Sci. 2005 Feb;60(2):224-31. doi: 10.1093/gerona/60.2.224. PMID 15814867
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] Vereeck L, Wuyts F, Truijen S, Van de Heyning P. Clinical assessment of balance: normative data, and gender and age effects. Int J Audiol. 2008 Feb;47(2):67-75. doi: 10.1080/14992020701689688. PMID 18236239
- [Derived] Shani P, Raeesi K, Walter E, Lewis K, Wang W, Cohen L, Yeh GY, Lengacher CA, Wayne PM. Qigong mind-body program for caregivers of cancer patients: design of a pilot three-arm randomized clinical trial. Pilot Feasibility Stud. 2021 Mar 19;7(1):73. doi: 10.1186/s40814-021-00793-4. PMID 33741070

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04019301/Prot_SAP_000.pdf